CLINICAL TRIAL: NCT01813890
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy and Safety of Tapentadol Immediate-Release Formulation in the Treatment of Acute Pain From Bunionectomy
Brief Title: A Study to Evaluate the Effectiveness and Safety of Tapentadol (CG5503) in the Treatment of Acute Pain From Bunionectomy Compared With Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Collaborators: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR101093; R331333PAI3035 (Other: Janssen-Cilag International NV)
Record Dates: First submitted 2013-03-15; First posted 2013-03-19 (Estimated); Results first posted 2015-01-09 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2014-12

CONDITIONS: Hallux Valgus
Keywords: Bunionectomy; Acute pain; Post-operative pain; Tapentadol IR; Analgesia; Hallux valgus
MeSH Terms: conditions — Hallux Valgus; Acute Pain; Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tapentadol IR 50 mg (Experimental)
  Interventions: Drug: Tapentadol IR 50 mg
- Tapentadol IR 75 mg (Experimental)
  Interventions: Drug: Tapentadol IR 75 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tapentadol IR 50 mg — Tapentadol IR 50 mg will be administered as a single oral dose once every 4 to 6 hours, during the double blind treatment period.
  Arms: Tapentadol IR 50 mg
Drug: Tapentadol IR 75 mg — Tapentadol IR 75 mg will be administered as a single oral dose once every 4 to 6 hours, during the double blind treatment period.
  Arms: Tapentadol IR 75 mg
Drug: Placebo — Placebo will be administered as a single oral dose once every 4 to 6 hours, during the double blind treatment period.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the analgesic efficacy and safety of tapentadol immediate-release (IR [CG5503]) for use in the relief of moderate to severe acute pain, compared with placebo, in adult Taiwanese patients with acute pain following bunionectomy.

DETAILED DESCRIPTION:
Patients undergoing bunionectomy (a surgical procedure to remove a bunion, an enlargement of the joint at the base of the big toe comprised of bone and soft tissue) often experience moderate to severe acute pain post-surgery. Normally such pain is controlled when patients receive repeated doses of opioid analgesics. Tapentadol (CG5503) is a newly synthesized opioid drug acting as a centrally acting analgesic like opioid analgesics but has a different mode of action. This study, a randomized (patients are assigned different treatments based on chance), double-blind (neither investigator nor patient knows which treatment the patient receives), placebo-controlled (placebo is an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial), parallel-group (each group of patients will be treated at the same time), multicenter study (the study is performed at more than one clinic) is designed to evaluate the effectiveness (level of pain control) and safety (side effects) of tapentadol immediate-release (IR) 50 mg or 75 mg versus placebo. The study will consist of a screening phase, during which the patients will be evaluated for study entry (Days -28 to -2) followed by the surgical period (Day -1) during which the bunionectomy will be performed and which will start with the first surgical incision and continues until termination of the popliteal sciatic block (PSB) infusion. During the qualification period (Day 1) which starts after termination of the post-operative continuous PSB infusion, patients will be evaluated for entry in the double blind treatment phase. Patients will be randomly assigned to one of three treatment groups to receive either 50 mg tapentadol IR, 75 mg tapentadol IR or a placebo if their PI is equal to or greater than 4 on a 0-10 numerical rating scale. The inpatient double-blind treatment period will be 72 hours in duration and will include a final end-of-double-blind evaluation (on Day 4, i.e., 72 hours after the administration of the first dose) for all patients. Any patient requiring analgesia for pain relief in addition to study drug during the double-blind treatment period will be discontinued from the study due to lack of efficacy. All patients who discontinue for lack of efficacy will complete pain assessments and the Patient Global Impression of Change (PGIC) before receiving rescue medication. Pain intensity and pain relief will be periodically assessed during the treatment period using rating scales. Safety evaluations include monitoring of adverse events, physical examinations, and clinical laboratory tests. The study length, including the screening period, will be up to a maximum duration of 32 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be undergoing primary unilateral first metatarsal bunionectomy that includes a distal Chevron osteotomy only, with or without the Akin procedure
* Patients must be healthy or medically stable on the basis of clinical laboratory tests performed at screening
* Women must be postmenopausal, surgically sterile, abstinent, or practicing or agree to practice an effective method of birth control and have a negative serum pregnancy test at screening and a negative urine pregnancy test before surgery
* If a male, must use an approved method of birth control and does not donate sperm from the day of study drug administration until 3 months afterwards
* Qualifying baseline Pain Intensity must be rated as greater than or equal to 4 on an 11-point (0 to 10) PI NRS, recorded within 30 minutes before randomization, no earlier than 10 hours after the first surgical incision and within 9 hours after termination of the continuous Popliteal Sciatic Block (PSB) infusion Exclusion Criteria: - History of seizure disorder or epilepsy, severe traumatic brain injury, episode(s) of unconsciousness of more than 24 hours duration, malignancy in the past 2 years with the exception of successfully treated basal cell carcinoma
* Mild or moderate traumatic brain injury, stroke, transient ischemic attack, or brain neoplasm within 1 year of screening
* Renal insufficiency, impaired hepatic function
* Use of anticonvulsants, monoamine oxidase inhibitors (MAOIs), tricyclic antidepressants (TCAs), neuroleptics, serotonin norepinephrine reuptake inhibitors (SNRIs), selective serotonin reuptake inhibitors (SSRIs) or triptans

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (3):
- Taiwan (3):
  - Kaohsiung City
  - Taipei
  - Taoyuan District

REFERENCES:
- [Derived] Chen YJ, Chiang CC, Huang PJ, Huang J, Karcher K, Li H. Tapentadol immediate-release for acute postbunionectomy pain: a phase 3, randomized, double-blind, placebo-controlled, parallel-group study in Taiwan. Curr Med Res Opin. 2015 Nov;31(11):2001-9. doi: 10.1185/03007995.2015.1082992. Epub 2015 Sep 21. PMID 26293513

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 11 January 2013 to 12 January 2014. Participants were recruited at 3 study centers in Taiwan.
Groups:
- Placebo: Placebo matched to tapentadol tablet administered orally,every 4 to 6 hours for 3 days.
- Tapentadol IR 50 mg: Tapentadol 50 milligram (mg) immediate release (IR) tablet administered orally, every 4 to 6 hours for 3 days.
- Tapentadol IR 75 mg: Tapentadol 75 mg IR tablet administered orally, every 4 to 6 hours for 3 days.
Period: Overall Study
Arm/Group | Placebo | Tapentadol IR 50 mg | Tapentadol IR 75 mg
Started | 20 | 21 | 19
Completed | 11 | 17 | 13
Not Completed | 9 | 4 | 6
Not completed — Adverse Event | 0 | 3 | 4
Not completed — Lack of Efficacy | 9 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tapentadol IR 50 mg | Tapentadol IR 75 mg | Total
Number analyzed (Participants) | 20 | 21 | 19 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (14.98) | 42.3 (14.27) | 43.3 (11.81) | 43.3 (13.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 18 | 58
  Male | 1 | 0 | 1 | 2
Age Customized [Number; unit: participants]
  Less than (<) 65 years | 18 | 20 | 18 | 56
  Greater than or equal (>=) to 65 years | 2 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Difference (SPID) Over 48 Hours
Description: Pain Intensity (PI) was assessed on an 11-point numerical rating scale from 0=no pain to 10=pain as bad as you can imagine. PID was the difference between baseline PI (prior to the first dose) and current PI at assessment. SPID was calculated as the time-weighted Sum of PID scores over 48 hours. Total score ranges from -480 (worst) to 480 (best) for SPID48. A higher value of SPID indicates greater pain relief.
Time Frame: 48 hours
Population: Intent-to-treat (ITT) analysis set, which included all randomly assigned participants with at least 1 dose of study medication. Last-observation-carried-forward imputation method was used for missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tapentadol IR 50 mg | Tapentadol IR 75 mg
Number analyzed (Participants) | 20 | 21 | 19
units on a scale | 50.8 (158.52) | 168.4 (84.50) | 194.9 (131.13)
Statistical Analysis 1: Comparison: Placebo vs Tapentadol IR 50 mg; Based on participant availability in Taiwan it was expected that 60 subjects (20 per group) would be enrolled. In consultation with the Taiwan health authority, the overall two-sided significance level was set at 0.20 (0.10 for each tapentadol versus placebo comparison). Assuming a standard deviation of 134.4, this sample size would provide 71.5% power to detect a between-group difference in SPID48 of 94.1 and 81.2% power to detect a between-group difference of 107.52; Test type: Superiority or Other; p = 0.006, ANCOVA — P-value adjusted for multiple treatment group comparisons using the Hochberg method; ANCOVA model with treatment group and center as factors and baseline pain intensity as covariate; Mean Difference (Net) = 105.61, 95% CI 2-sided [32.0 to 179.2] — Difference is SPID48 in tapentadol IR group minus SPID48 in placebo group
Statistical Analysis 2: Comparison: Placebo vs Tapentadol IR 75 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.004, ANCOVA — P-value adjusted for multiple treatment group comparisons using the Hochberg method; ANCOVA model with treatment group and center as factors and baseline pain intensity as covariate; Median Difference (Net) = 126.58, 95% CI 2-sided [49.5 to 203.7] — Difference is SPID48 in tapentadol IR group minus SPID48 in placebo group

2. Secondary Outcome: Time to First Rescue Medication Use
Description: Rescue medication was defined as any analgesic medication used for participants discontinued due to lack of efficacy (including those started at time of discontinuation) or analgesic medication used during the double-blind period for completed participants.
Time Frame: up to 48 hours
Population: ITT analysis set, which included all randomly assigned participants with at least 1 dose of study medication.
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Placebo | Tapentadol IR 50 mg | Tapentadol IR 75 mg
Number analyzed (Participants) | 20 | 21 | 19
Hours | NA (84.50) [8.1 to NA] — The median time to the first rescue medication could not be calculated for the treatment group because only 50 percent of participants used rescue medication. | NA (131.13) [NA to NA] — The median time to the first rescue medication could not be calculated for the treatment group because less than 50 percent (1 [4.8 percent]) of participants used rescue medication. | NA (158.52) [NA to NA] — The median time to the first rescue medication could not be calculated for the treatment group because less than 50 percent (2 [10.5 percent]) of participants used rescue medication.

3. Secondary Outcome: Response Rate for 30 Percent or Greater Reduction in Pain Intensity at 12, 24, 48 and 72 Hours
Description: Response rate was defined as the percentage of participants with a 30 percent or greater reduction in pain intensity from baseline to 12, 24, 48, and 72 hours. Pain intensity was assessed on a 11-point numerical rating scale from 0=no pain to 10=pain as bad as you can imagine. Participants with no assessment at the given time point, who used an analgesic medication prior to the time point, or who had worse pain intensity at the time point compared to baseline were assigned a percent reduction of 0 percent.
Time Frame: 12, 24, 48 and 72 hours
Population: ITT analysis set, which included all randomly assigned participants with at least 1 dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Tapentadol IR 50 mg | Tapentadol IR 75 mg
Number analyzed (Participants) | 20 | 21 | 19
Percentage of Participants
  12 hours | 35.0 | 66.7 | 73.7
  24 hours | 40.0 | 66.7 | 73.7
  48 hours | 45.0 | 81.0 | 68.4
  72 hours | 45.0 | 81.0 | 68.4

4. Secondary Outcome: Response Rate for 50 Percent or Greater Reduction in Pain Intensity at 12, 24, 48 and 72 Hours
Description: Response rate was defined as the percentage of participants with a 50 percent or greater reduction in pain intensity from baseline to 12, 24, 48, and 72 hours. Pain intensity was assessed on a 11-point numerical rating scale from 0=no pain to 10=pain as bad as you can imagine. Participants with no assessment at the given time point, who used an analgesic medication prior to the time point, or who had worse pain intensity at the time point compared to baseline were assigned a percent reduction of 0 percent.
Time Frame: 12, 24, 48 and 72 hours
Population: ITT analysis set, which included all randomly assigned participants with at least 1 dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Tapentadol IR 50 mg | Tapentadol IR 75 mg
Number analyzed (Participants) | 20 | 21 | 19
Percentage of Participants
  12 hours | 20.0 | 42.9 | 57.9
  24 hours | 35.0 | 61.9 | 73.7
  48 hours | 40.0 | 76.2 | 68.4
  72 hours | 45.0 | 81.0 | 68.4

5. Secondary Outcome: Sum of Pain Intensity Differences (SPID) Over 12, 24 and 72 Hours
Description: Pain Intensity (PI) was assessed on an 11-point numerical rating scale from 0=no pain to 10=pain as bad as you can imagine. PID was the difference between baseline PI (prior to the first dose) and current PI at assessment. SPID was calculated as the time-weighted Sum of PID scores over 12, 24, and 72 hours. Total score ranges from -120 (worst) to 120 (best) for SPID12, -240 (worst) to 240 (best) for SPID24, -720 (worst) to 720 (best) for SPID72. A higher value of SPID indicates greater pain relief.
Time Frame: 12, 24 and 72 hours
Population: ITT analysis set, which included all randomly assigned participants with at least 1 dose of study medication. Last-observation-carried-forward imputation method was used for missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tapentadol IR 50 mg | Tapentadol IR 75 mg
Number analyzed (Participants) | 20 | 21 | 19
units on a scale
  12 hours | 7.6 (32.22) | 30.3 (17.24) | 34.7 (25.70)
  24 hours | 16.7 (69.37) | 67.5 (40.90) | 82.0 (57.65)
  72 hours | 91.6 (252.89) | 281.3 (129.48) | 316.1 (206.81)

6. Secondary Outcome: Total Pain Relief (TOTPAR) Over 12, 24, 48, and 72 Hours
Description: Participants rated pain relief on 5-point categorical scale of 0-4 (0=none, 1=A little, 2=Some, 3=A lot, 4=Complete). Total Pain Relief (TOTPAR) was calculated as the time-weighted sum of pain relief scores up to Hour 12, 24, 48, and 72. Total score ranges from 0 (worst) to 48 (best) for TOTPAR12, 0 (worst) to 96 (best) for TOTPAR24, 0 (worst) to 192 (best) for TOTPAR48, and 0 (worst) to 288 (best) for TOTPAR72. A higher value of TOTPAR indicated greater pain relief.
Time Frame: 12, 24, 48, and 72 hours
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tapentadol IR 50 mg | Tapentadol IR 75 mg
Number analyzed (Participants) | 20 | 21 | 19
units on a scale
  12 hours | 13.0 (11.29) | 22.5 (10.27) | 24.4 (10.33)
  24 hours | 28.0 (24.50) | 48.2 (22.07) | 54.1 (20.47)
  48 hours | 68.2 (62.26) | 115.6 (45.06) | 123.5 (49.99)
  72 hours | 112.6 (103.19) | 187.3 (68.03) | 194.1 (74.63)

7. Secondary Outcome: Sum of Pain Relief and Pain Intensity Differences (SPRID) Over 12, 24, 48, and 72 Hours
Description: Participants rated pain relief on 5-point categorical scale of 0-4 (0=none, 1=A little, 2=Some, 3=A lot, 4=Complete). Pain Intensity (PI) was assessed on an 11-point numerical rating scale from 0=no pain to 10=pain as bad as you can imagine. PID was the difference between baseline PI (prior to the first dose) and current PI at assessment. PRID is the sum of pain relief and PID at the same assessment time. SPRID was calculated as the time-weighted Sum of PRID scores over 12, 24, 48, and 72 hours. Total score ranges from -120 (worst) to 168 (best) for SPRID12, -240 (worst) to 336 (best) for SPRID24, -480 (worst) to 672 (best) for SPRID48, and -720 (worst) to 1008 (best) for SPRID72. A higher value of SPRID indicates greater pain relief.
Time Frame: 12, 24, 48 and 72 hours
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tapentadol IR 50 mg | Tapentadol IR 75 mg
Number analyzed (Participants) | 20 | 21 | 19
units on a scale
  12 hours | 20.7 (41.51) | 52.8 (25.66) | 59.1 (33.20)
  24 hours | 44.7 (90.14) | 115.7 (59.74) | 136.0 (72.59)
  48 hours | 119.1 (214.14) | 284.0 (122.07) | 318.4 (171.50)
  72 hours | 204.3 (346.52) | 468.6 (185.43) | 510.2 (268.96)

8. Secondary Outcome: Patient Global Impression of Change (PGI-C) Score at 72 Hours
Description: The PGI-C is a 7-point scale that requires the participants to assess how much their illness has improved or worsened relative to a baseline state at the beginning of the intervention. The response options are: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; and 7=very much worse. Higher scores indicate worsening.
Time Frame: Baseline (Day 1) and 72 hours
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tapentadol IR 50 mg | Tapentadol IR 75 mg
Number analyzed (Participants) | 20 | 21 | 19
Percentage of participants
  Very Much Improved | 40.0 | 71.4 | 73.7
  Much Improved | 10.0 | 14.3 | 5.3
  Minimally Improved | 5.0 | 9.5 | 10.5
  No Change | 20.0 | 4.8 | 0.0
  Minimally Worse | 0.0 | 0.0 | 0.0
  Much Worse | 0.0 | 0.0 | 0.0
  Very Much Worse | 25.0 | 0.0 | 10.5

ADVERSE EVENTS:
Arm/Group | Placebo | Tapentadol IR 50 mg | Tapentadol IR 75 mg
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 3/20 | 19/21 | 18/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=20) | Tapentadol IR 50 mg (N=21) | Tapentadol IR 75 mg (N=19)
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 7 | 8
Vomiting (Gastrointestinal disorders) | 0 | 4 | 10
Chest discomfort (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 3 | 2
Wound complication (Injury, poisoning and procedural complications) | 0 | 2 | 0
Dizziness (Nervous system disorders) | 1 | 14 | 16
Headache (Nervous system disorders) | 1 | 3 | 2
Somnolence (Nervous system disorders) | 0 | 3 | 2
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days